CLINICAL TRIAL: NCT01810289
Title: The "START" (a Streamlined ART Initiation Strategy) Study
Acronym: START-ART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: START-ART
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: HIV
Keywords: HIV, ART, CD4

STUDY DESIGN:
Intervention Model Description: Clinic level stepped wedge design where each clinic has an amount of time in the pre-intervention or standard of care condition and then crosses over in the intervention condition
Oversight: Data Monitoring Committee: No

ARMS (2):
- MJAP Clinics Intervention (Experimental): START intervention. This is a stepped wedge design so each clinic will experience both conditions.
  Interventions: Behavioral: START
- MJAP Clinics Pre-Intervention (No Intervention): Standard of care. This is a stepped wedge design so each clinic will experience both conditions.

INTERVENTIONS:
Behavioral: START — INTERVENTION: START is clinic-level (not individual-patient) intervention to catalyze the process of ART initiation among HIV-infected adults who meet CD4-based criteria for combination ART (e.g., adults with a CD4 T cell level < 350/ul). The three START components are: (1) real-time point-of-care CD4 testing using the Alere PIMA platform to ascertain treatment eligibility in real time at first presentation to care, (2)targeted knowledge transfer(i.e., dissemination) of recent scientific evidence regarding effects rapid ART initiation on survival to front line health care workers; and 3)feedback and reporting to clinic and providers. There three components represent empirically validated steps in the PRECEED implementation model.
  This intervention will be implemented at all Makerere Joint AIDS Program (MJAP) clinics in Kampala and Mbarara districts in a step-wedge design.
  Arms: MJAP Clinics Intervention

SUMMARY:
START is clinic-level (not individual-patient) intervention to catalyze the process of ART initiation among HIV-infected adults who meet CD4-based criteria for combination ART (e.g., adults with a CD4 T cell level < 350/ul). The three START components are: (1) real-time point-of-care CD4 testing using the Alere PIMA platform to ascertain treatment eligibility in real time at first presentation to care, (2) targeted knowledge transfer (i.e., dissemination) of recent scientific evidence regarding effects rapid ART initiation on survival to front line health care workers; and 3) feedback and reporting to clinic and providers. There three components represent empirically validated steps in the PRECEED implementation model.

DETAILED DESCRIPTION:
RATIONALE: In Africa, up to a 50-75% of HIV-infected, adults fail to initiate (FTI) ART or encounter delays of months even after eligibility through CD4+ T-cell testing or clinical criteria are established. Recent randomized trials including ACTG Protocol 5164, ACTG 5221, CAMELIA and SAPIT have demonstrated that delays of even weeks in ART initiation increases mortality among patients presenting with active opportunistic infections. Even among those without active infections, mortality among untreated persons with a CD4 < 350 approaches 15/100 person-years - a large proportion of which should be avoidable in patients who have presented to care. New dissemination and implementation strategies that are generalizable across resource-limited settings are needed to address FTI and make the public health approach more effective. The overall goal of the multi-component START strategy is to initiate the greatest number of eligible patients in the shortest amount of time possible, while maintaining safety, efficacy and cost effectiveness.

HYPOTHESIS: The START intervention, a combined intervention using provider education, novel technology and reinforcing feedback, will increase the rapidity and completeness of ART initiation.

INTERVENTION: START is clinic-level (not individual-patient) intervention to catalyze the process of ART initiation among HIV-infected adults who meet CD4-based criteria for combination ART (e.g., adults with a CD4 T cell level < 350/ul). The three START components are: (1) real-time point-of-care CD4 testing using the Alere PIMA platform to ascertain treatment eligibility in real time at first presentation to care, (2) targeted knowledge transfer (i.e., dissemination) of recent scientific evidence regarding effects rapid ART initiation on survival to front line health care workers; and 3) feedback and reporting to clinic and providers. There three components represent empirically validated steps in the PRECEED implementation model.

STUDY DESIGN: A cluster-randomized, step-wedge trail of 20 clinics operated by the Makerere Joint AIDS Program. Four clinic sites will be randomly assigned to the START at 6-month intervals between month six and 24 during the three-year trial.

PRIMARY OBJECTIVE

1. Evaluate the programmatic change of START on the cumulative incidence of ART initiation 14 days after first clinical eligibility for ART in treatment eligible HIV-infected patients receiving care under routine program conditions in a large, multi-site, HIV care program in Uganda.

SECONDARY OBJECTIVES

1. Evaluate the effect of START on the incidence of mortality in treatment-eligible, HIV-infected patients.
2. Evaluate the effect of START on plasma HIV RNA levels one year after treatment eligibility in HIV-infected patients presenting to care in a multi-site, HIV care program.
3. Evaluate the effect of START on the incidence of vertical transmission in all treatment-eligible, HIV-infected women.
4. Evaluate the effect of START on retention among ART-eligible, HIV-infected patients in the study sites.
5. To assess the cost-effectiveness of the START intervention.
6. To evaluate adaptation of START intervention into clinical care through qualitative analysis of counseling interactions and limited interviews with counselors and patients regarding their experience of counseling and identification of content of current counseling activities and how this changes over time.

OUTCOMES: The primary outcome of the study is ART initiation. Secondary outcomes are all-cause mortality, plasma HIV RNA at one year after clinic presentation, vertical transmission events and cost-effectiveness measures.

ANALYTIC PLAN:

Primary analysis for primary outcome:

We will treat the outcome as binary, in which we consider patients as either initiating ARV by 14 days or not. In other words, the outcome of ART start within 14 days or less is met if the start is by 14 days inclusive (<=14 days), otherwise the outcome is not met. Patients with less than 14 days of observation time before cross-over or end of study database closure will not be analyzed. This means that even if a patient initiates ART but has less than 14 days of possible observation time, that event will not be counted. Also, deaths prior to ARV initiation are considered non-initiations. The analysis will use a mixed effect logistic regression model (meglm in Stata 14.0) with a Normal random effect for site and a fixed effect for intervention. Marginal proportions will under intervention and control be calculated using the "margins" command in Stata. We will represent the effect as a risk ratio of marginal proportions.

Secondary sensitivity analyses for primary outcome

1. We will adjust the primary analysis for calendar time specified as a restricted cubic spline.
2. We will restrict analyses to the incidently eligible population.
3. We will perform an analysis including all observation time censoring those with less than 14 days of observation due to database closure or cross-over.
4. We will carry out an analysis in which we estimate the effect of crossing into the intervention condition among patients who are eligible but who had not started ART at the time clinics changed from control to intervention through introduction of a time-varying covariate representing cross over date in a multivariable regression model.

ELIGIBILITY:
Inclusion Criteria:

* All MJAP-supported clinics in Kampala and Mbarara Districts

Exclusion Criteria:

* None.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12024 (Actual)
Dates: Start 2013-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane V Havlir, MD, Principal Investigator — University of California, San Francisco; Moses Kamya, MB.Ch.B, Principal Investigator — Makerere University; Elvin Geng, MD, MPH, Principal Investigator — University of California, San Francisco

REFERENCES:
- [Result] Amanyire G, Semitala FC, Namusobya J, Katuramu R, Kampiire L, Wallenta J, Charlebois E, Camlin C, Kahn J, Chang W, Glidden D, Kamya M, Havlir D, Geng E. Effects of a multicomponent intervention to streamline initiation of antiretroviral therapy in Africa: a stepped-wedge cluster-randomised trial. Lancet HIV. 2016 Nov;3(11):e539-e548. doi: 10.1016/S2352-3018(16)30090-X. Epub 2016 Aug 27. PMID 27658873
- [Derived] Hodgson S, Griffin TJ, Reilly C, Harvey S, Witthuhn BA, Sandri BJ, Kunisaki KM, Wendt CH. Plasma sphingolipids in HIV-associated chronic obstructive pulmonary disease. BMJ Open Respir Res. 2017 Apr 3;4(1):e000180. doi: 10.1136/bmjresp-2017-000180. eCollection 2017. PMID 28409005

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-intervention: This study is stepped-wedge in design, therefore each clinic experienced a period of time before the intervention rolled out and then a time period after the intervention rolled out. Each clinic contributes time to both conditions. In the pre-intervention condition the clinic is using the standard of care.
- Post-intervention: This study is stepped-wedge in design, therefore each clinic experienced a period of time before the intervention rolled out and then a time period after the intervention rolled out. Each clinic contributes time to both conditions. In the intervention condition ("post-intervention") the clinics have received the intervention - training, ongoing feedback, as well as the point of care CD4 (PIMA) machine.
Period: Overall Study
Arm/Group | Pre-intervention | Post-intervention
Started | 7277 | 4747
Completed | 7277 | 4747
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A patient is considered in pre-intervention group (control) if becoming eligible for ART initiation during a time period prior to the roll out of the intervention at the clinic. A patient is grouped into the intervention if becoming eligible for ART initiation during a time period after the roll out of the intervention at the clinic.
Groups:
- Pre-intervention; Post-intervention: This study is stepped-wedge in design, so each clinic experienced a period of time before the intervention rolled out and then a time period after the intervention rolled out. Each clinic contributes time to both conditions.
- Total: Total of all reporting groups
Arm/Group | Pre-intervention | Post-intervention | Total
Number analyzed (Participants) | 7277 | 4747 | 12024
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31 [26 to 38] | 30 [25 to 37] | 31 [26 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4715 | 2830 | 7545
  Male | 2562 | 1917 | 4479

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of ART Initiation 14 Days After Clinical Eligibility in Treatment Eligible HIV-infected Patients
Description: Patients may be ART eligible at the start of the study or become ART eligible for the first time in the 3 year time frame.
Time Frame: 14 days
Population: Persons who did have the opportunity for 14 days of follow up were excluded from these analyses.
Measure: Number; unit: participants
Groups:
- Pre-intervention: This study is stepped-wedge in design, so each clinic experienced a period of time before the intervention rolled out and then a time period after the intervention rolled out. Each clinic contributes time to both conditions. Clinics in the pre-intervention condition are giving the standard of care.
- Post-intervention: This study is stepped-wedge in design, so each clinic experienced a period of time before the intervention rolled out and then a time period after the intervention rolled out. Each clinic contributes time to both conditions. Clinics in the intervention ("post-intervention") have experienced training, ongoing feedback and have the PIMA machine.
Arm/Group | Pre-intervention | Post-intervention
Number analyzed (Participants) | 7066 | 4747
participants | 2585 | 3753

2. Secondary Outcome: Incidence of Mortality in Treatment-eligible, HIV-infected Patients.
Description: We ascertained mortality in the subgroup of those selected for HIV RNA assessment. Vital status is not reliably reported in program data. Assessment was 1 year after ART eligibility.
Time Frame: 1 years
Population: Mortality information is not systematically measured in the program data. We assessed this outcome in the subgroup selected for HIV RNA.
Measure: Number; unit: percentage of reported deaths
Arm/Group | Pre-intervention | Post-intervention
Number analyzed (Participants) | 199 | 208
percentage of reported deaths | 3 | 2

3. Secondary Outcome: Retention in HIV Care Among Treatment-eligible, HIV-infected Patients.
Description: Retention was operationalized as the proportion of appointments made within 7 days within one year after ART eligibility.
Time Frame: 1 years
Population: Retention was assess among all in the study
Measure: Number; unit: percentage of appointments made
Units Other Than Participants: Appointments
Arm/Group | Pre-intervention | Post-intervention
Number analyzed (Participants) | 7277 | 4747
Number analyzed (Appointments) | 25920 | 15241
percentage of appointments made | 84 | 84

4. Secondary Outcome: HIV RNA Levels Among Treatment-eligible, HIV-infected Patients One Year Following ART Eligibility
Description: Due to financial constraints, HIV RNA was measured in a random sample of patients to asses virologic suppression.
Time Frame: 1 year
Population: A total of 437 (217 in control + 220 in intervention) patients were selected for blood samples. We did two analyses, one treating missing as failure and another using inverse probability weighting to address missing outcomes. The primary reported here is missing as failure.
Measure: Number; unit: percentage of participants
Arm/Group | Pre-intervention | Post-intervention
Number analyzed (Participants) | 217 | 220
percentage of participants | 58 | 66

5. Secondary Outcome: Incidence of Vertical Transmission in All HIV-infected Women Who Are Treatment-eligible During the Study Period.
Time Frame: 3 years
Population: Linking children to mothers in a systematic way was unattainable in these program data. We were unable to ascertain this outcome.
Arm/Group | Pre-intervention | Post-intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Pre-intervention | Post-intervention
Serious Adverse Events (participants affected / at risk) | 0/7277 | 0/4747
Other Adverse Events (participants affected / at risk) | 0/7277 | 0/4747

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No